CLINICAL TRIAL: NCT04323189
Title: Effects of Sitagliptin in Individuals With Genetically Decreased DPP4
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jessica R.Wilson, MD, MS, Instructor in Medicine, Division of Endocrinology, Diabetes, and Metabolism, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 834482
Record Dates: First submitted 2019-03-25; First posted 2020-03-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Genetics Disease; Type2 Diabetes; Heart Failure
Keywords: genetics; sitagliptin; DPP4 inhibition; heart failure; type 2 diabetes
MeSH Terms: conditions — Genetic Diseases, Inborn; Heart Failure; Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Intervention Model Description: blinded 2:2 crossover, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither subjects, nor the investigator or key study personnel will know drug randomization until after data analyses are completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crossover AB (Other): Subjects in arm A will first receive placebo daily for 7 days in the first intervention followed by sitagliptin 100mg/d for 7 days in the crossover intervention.
  Interventions: Drug: Sitagliptin 100mg; Drug: Placebo Oral Tablet
- Crossover BA (Other): Subjects in arm B will first receive sitagliptin 100mg/d for 7 days in the first intervention followed by placebo for 7 days in the crossover intervention.
  Interventions: Drug: Sitagliptin 100mg; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sitagliptin 100mg — Sitagliptin will be administered daily for 7 days, with a study day on day 7.
  Other Names: Januvia
Drug: Placebo Oral Tablet — Placebo will be administered daily for 7 days, with a study day on day 7.

SUMMARY:
This is a pilot clinical trial to test the hypothesis that during sitagliptin (DPP4 inhibitor), individuals heterozygous for DPP4 loss of function variants will have a reduction in DPP4 activity and antigen, lower glucose after a mixed meal, and higher levels of intact DPP4 substrates compared to during placebo and compared to matched controls.

DETAILED DESCRIPTION:
Participants of this pilot clinical trial will be randomized in a blinded 2:2 crossover manner to receive placebo and sitagliptin 100 mg/d (DPP4 inhibitor), in random order. Subjects will receive each intervention for seven days, with a study day on day 7. Each intervention will be separated by a 4-week washout period. Each subject will have up to four separate visits: 1) DXA, echocardiogram, 2) cardiac MRI, 3) mixed meal during placebo, 4) mixed meal during sitagliptin.

The study will include 10 cases (heterozygous for DPP4 loss of function variant) and 10 controls.

ELIGIBILITY:
Inclusion Criteria:

* Participant of the Penn Medicine Biobank who is willing to be recontacted to participate in future research.
* Cases are defined as adults 18-70 years with likely decreased DPP4.
* Controls are defined as adults who are matched to cases by: age, gender, race, BMI, hypertension status, diabetes status, renal function, and medication use that may affect outcomes of interest.

Exclusion Criteria:

* The study will exclude volunteers with any significant medical conditions that may interfere with study participation, data interpretation, or pose safety risk(s) to the subject.
* Recent hospitalization or acute illness such as infection within the past two weeks
* Pregnancy
* Use of insulin
* Use of a GLP-1 agonist or DPP4 inhibitor medication
* Use of oral diabetes agents other than metformin unless matched with controls
* Type 1 diabetes
* Chronic steroid use or use within the last 30 days
* Significant liver disease including liver enzymes >3 x upper limit of normal range
* Renal dysfunction defined as eGFR< 50mL/min/1.73m2
* Significant cardiac disease such as heart transplantation
* Significant gastrointestinal conditions that may interfere with drug absorption or GLP-1 release including bariatric surgery
* Significant hematologic disease such as hematocrit <35%
* Use of chronic anticoagulation
* Severe pulmonary disease
* Severe neurologic or psychiatric disease
* Inability to comprehend study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Dipeptidyl peptidase 4 (DPP4) | during study days 1 and 2
  DPP4 activity and antigen concentration

SECONDARY OUTCOMES:
Glucose Area Under the Curve | Before the meal and for 4 hours after (t=-15 through t=240 min) on study days 1 and 2
  Glucose will be measured before after the mixed meal during sitagliptin and placebo. Area under the curve will be calculated based on at least 10 time points after the meal.
Disposition index | Calculated from samples collected before the meal and for 4 hours after (t=-15 through t=240 min) on study days 1 and 2
  Disposition index will be calculated from insulin sensitivity and insulin secretion. These variables will be computed using mathematical modeling of insulin and c-peptide. We will collect insulin and c-peptide at least 10 time points after the meal.
Mean blood pressure | Before the meal and for 4 hours after (t=-15 through t=240 min) on study days 1 and 2
  Measured via an automated blood pressure cuff approximately every 15 minutes
Glucagon-like peptide-1 (GLP-1) | Before the meal and for 4 hours after (t=-15 through t=240 min) on study days 1 and 2
  This is released in response to a meal and rapidly degraded by DPP4. We will collect samples for at least six time points after the meal.
CD26 | Before the meal or at baseline (t=-15 or -1 min) on study days 1 and 2
  CD26 is DPP4 on T cells and monocytes.
Surrogate markers of lipolysis | Before the meal and for 4 hours after (t=-15 through t=240 min) on study days 1 and 2
  Triglycerides, free fatty acids; We will collect samples at least six time points after the meal.
Mean heart rate | Before the meal and for 4 hours after (t=-15 through t=240 min) on study days 1 and 2
  Measured via an automated blood pressure cuff approximately every 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Wilson, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be deidentified for outcomes of interest from this pilot study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified data will become available upon completion of the pilot study